CLINICAL TRIAL: NCT07291271
Title: Flow-controlled Ventilation During Percutaneous CT-guided Liver Tumor Ablation
Brief Title: Use of Flow-Controlled Ventilation During CT-Guided Percutaneous Liver Tumor Ablation
Acronym: EVOLVE
Status: Completed | Type: Observational
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, Hannah Schulz, Drs, MD., Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Other Study IDs: METc-number: 2024.0386
Record Dates: First submitted 2025-11-25; First posted 2025-12-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Ventilation; Ablation Techniques
Keywords: Flow controlled ventilation; Volume controlled ventilation; Liver tumor; Percutaneous ablation; CT-guided ablation
MeSH Terms: conditions — Respiratory Aspiration; Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Flow controlled ventilation: Patients recieving CT-guided percutaneous ablation, ventilated with flow controlled ventilation
  Interventions: Device: Flow controlled ventilation
- Volume controlled ventilation: Patients recieving CT-guided percutaneous ablation, ventilated with volume controlled ventilation

INTERVENTIONS:
Device: Flow controlled ventilation — Flow controlled ventilation will be investigated during CT-guided percutaneous ablation of liver tumors
  Groups: Flow controlled ventilation

SUMMARY:
Tumors in the liver can be treated using percutaneous ablation. At the Amsterdam UMC, this procedure is often performed under CT guidance by an interventional radiologist. The available ablation techniques include thermal ablation (microwave ablation (MWA) and radiofrequency ablation (RFA)) and non-thermal ablation (irreversible electroporation (IRE)). Thermal ablation is performed under general anesthesia or deep sedation, whereas non-thermal ablation is always performed under general anesthesia.

Flow-controlled ventilation (FCV) is a ventilation technique in which increased diaphragm stability is observed due to a continuous flow during both inspiration and expiration. This contrasts with volume- or pressure-controlled ventilation, where active inspiration is followed by passive expiration through an increase in pressure or flow, leading to greater diaphragm movement during the ventilation cycle. With volume- or pressure-controlled ventilation, diaphragm position fluctuates between inspiration and expiration, requiring temporary pauses in ventilation (apnea; allowing the diaphragm to become motionless) during ablation needle positioning.

During volume- or pressure-controlled ventilation and the associated apnea periods, increased formation of atelectasis is often observed. This results in changes in diaphragm position during and after each apnea, which can complicate accurate needle placement. With FCV, apnea is not necessary-the continuous flow results in minimal diaphragm excursion and can be maintained throughout the entire procedure without interruption.

Both ventilation modes are currently used during CT-guided percutaneous ablation of liver and pancreatic tumors. However, the choice of ventilation technique presently lies with the attending anesthesiologist. In practice, some anesthesiologists prefer volume- or pressure-controlled ventilation, as these are traditionally the most commonly used modes. Others opt for FCV due to its minimal effect on diaphragm excursion and its potentially beneficial effects on atelectasis formation and intraprocedural image quality.

Given the subdiaphragmatic location of both organs and the presence of critical surrounding structures that must be preserved during the procedure, interventional radiologists find FCV particularly advantageous. Moreover, continuous ventilation without apnea is preferred by anesthesiologists, as it avoids periods of reduced oxygenation.

FCV is an already approved ventilation technique at Amsterdam UMC and is used during percutaneous ablations, surgeries performed by ENT and pulmonary specialists, and in the intensive care unit for critically ill patients. Through this study, the investigators aim to evaluate the use of FCV as a ventilation technique during CT-guided percutaneous ablations of liver tumors and to compare it with volume- or pressure-controlled ventilation.

ELIGIBILITY:
Inclusion Criteria:

* Clinical indication for CT-guided percutaneous ablation of one or more liver tumours
* Approval for general anaesthesia

Exclusion Criteria:

* Procedures performed under procedural sedation
* Uncontrolled asthma, and (4) COPD classified as Global Initiative for Chronic Obstructive Lung Disease (GOLD) stage III or IV
* No signed informed consent form

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients eligible for CT-guided percutaneous ablation of liver tumors
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2024-08-20 (Actual); Primary Completion 2025-05-20 (Actual); Study Completion 2025-11-20 (Actual)

PRIMARY OUTCOMES:
Switch from flow controlled ventilation to volume controlled ventilation | During the CT-guided percutaneous ablation procedure
  Switch if deemed necessary by the anesthesiologist performing the ventilation.

SECONDARY OUTCOMES:
Image-based analyses | During the ablation procedure
  Comparison of diaphragm movement by segmenting the pulmonary bases in pre- and post-ablation images and assessment of intra-procedural atelectasis formation.
Modified five-point Surgical Rating Scale | Directly after the ablation procedure
  Completed by the interventional radiologist to assess the suitability of FCV for the procedure.
  Score can vary from 0-25, where 25 is the highest score.

CONTACTS AND LOCATIONS:
Locations (1):
- Amsterdam UMC, location VUmc, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided